CLINICAL TRIAL: NCT00424762
Title: Effect of Rosiglitazone Versus Placebo on Cardiovascular Performance and Myocardial Triglyceride
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry); Abbott RDx Cardiometabolic (Other)
Responsible Party: Principal Investigator, Darren McGuire, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GSK 102610
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Congestive Heart Failure; Cardiopulmonary exercise testing; intracellular cardiomyocyte triglycerides; thiazolidinedione; rosiglitazone; nuclear magnetic resonance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rosiglitazone (Experimental): 4mg titrated to 8mg daily
  Interventions: Drug: rosiglitazone
- Placebo (Placebo Comparator): blinded matching placebo treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rosiglitazone — 6 months of treatment of blinded study drug
  Other Names: Avandia
  Arms: rosiglitazone
Drug: placebo — blinded treatment with matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if rosiglitazone treatment improves integrated cardiovascular performance in patients at risk for congestive heart failure. A second aim of this study is to determine if treatment with rosiglitazone decreases intracellular (ectopic) triglyceride (TG) deposition in cardiomyocytes using nuclear magnetic resonance (NMR) techniques, and how changes in intra-myocardial lipid content relate to changes in cardiac structure and function.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD), including congestive heart failure (CHF), accounts for over 75% of deaths among patients with diabetes. Thus, it is imperative to rigorously evaluate existing and emerging hypoglycemic therapies with regard to their cardiovascular consequences. The thiazolidinedione (TZD) class of drugs, alone or in combination with other oral hypoglycemic medications or with insulin, has emerged as a safe and effective treatment of hyperglycemia in type 2 diabetes. Both in vitro and in vivo studies have revealed favorable pleiotropic effects of TZD on myocyte and ventricular structure and function. However, approximately 10% of patients taking TZDs develop peripheral edema and some patients have developed heart failure decompensation on the drug. These observations have led to a Food and Drug Administration (FDA) warning regarding the use of TZDs in patients with or at high risk of developing congestive heart failure (CHF). The exact effects of TZDs on integrated cardiovascular performance remain unclear. The primary hypothesis of this study is that TZD treatment improves integrated cardiovascular performance in patients at risk for CHF by improving both central (i.e. cardiac output) and peripheral (i.e. vascular resistance) function.

Recently, we have developed a sensitive, reproducible noninvasive assay to measure intra-cardiomyocyte fat, which varies widely in amount between individuals. The relationship between the amount of cardiomyocyte triglyceride accumulation and LV mass and function remains unclear. TZDs have been previously shown to be associated with decreases in the TG content of the liver and muscle. The secondary hypothesis being tested in this study is that TZD treatment improves cardiac function by decreasing intra-cardiac myocyte triglyceride content.

Comparisons:

* Peak oxygen uptake (VO2) during cardiopulmonary exercise testing in individuals randomized to rosiglitazone, compared to those on placebo.
* Amount of intra-myocardial triglycerides using NMR techniques in in individuals randomized to rosiglitazone, compared to those on placebo.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus (prior clinical diagnosis and current use of hypoglycemic medical therapy or by new diagnosis according to ADA criteria) with at least one of the following:

  * prior diagnosis of cardiovascular disease (CAD, MI, revascularization, CVA/TIA, carotid or peripheral arterial disease)
  * at least one additional CVD risk factor (smoking, hypertension, hypercholesterolemia, albuminuria, family history of premature CAD, or documented hsCRP>3)

Exclusion Criteria:

* treatment with a TZD within prior 6 months
* documented intolerance to TZD
* history or evidence of CHF
* AST/ALT>3X upper limits of normal
* creatinine >2.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren K McGuire, MD, MHSc, Principal Investigator — University of Texas Southwestern Medical Center; Darren K McGuire, M.D., MHSc, Study Chair — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] McGuire DK, See R, Abdullah SM, Snell PG, McGavock JM, Ayers CR, Szczepaniak LS. The effect of rosiglitazone on integrated cardiovascular performance, cardiac structure, function and myocardial triglyceride: trial design and rationale. Diab Vasc Dis Res. 2009 Jan;6(1):43-50. doi: 10.3132/dvdr.2009.009. PMID 19156629
- [Result] McGuire DK, Abdullah SM, See R, Snell PG, McGavock J, Szczepaniak LS, Ayers CR, Drazner MH, Khera A, de Lemos JA. Randomized comparison of the effects of rosiglitazone vs. placebo on peak integrated cardiovascular performance, cardiac structure, and function. Eur Heart J. 2010 Sep;31(18):2262-70. doi: 10.1093/eurheartj/ehq228. Epub 2010 Jul 2. PMID 20601395
- [Derived] Jarvie JL, Pandey A, Ayers CR, McGavock JM, Senechal M, Berry JD, Patel KV, McGuire DK. Aerobic Fitness and Adherence to Guideline-Recommended Minimum Physical Activity Among Ambulatory Patients With Type 2 Diabetes Mellitus. Diabetes Care. 2019 Jul;42(7):1333-1339. doi: 10.2337/dc18-2634. Epub 2019 May 21. PMID 31221698
- [Derived] McGavock J, Szczepaniak LS, Ayers CR, Abdullah SM, See R, Gore MO, Drazner MH, de Lemos JA, McGuire DK. The effects of rosiglitazone on myocardial triglyceride content in patients with type 2 diabetes: a randomised, placebo-controlled trial. Diab Vasc Dis Res. 2012 Apr;9(2):131-7. doi: 10.1177/1479164111428628. Epub 2011 Nov 8. PMID 22067724
- [Derived] Narang N, Armstead SI, Stream A, Abdullah SM, See R, Snell PG, McGavock J, Ayers CR, Gore MO, Khera A, de Lemos JA, McGuire DK. Assessment of cardiac structure and function in patients without and with peripheral oedema during rosiglitazone treatment. Diab Vasc Dis Res. 2011 Apr;8(2):101-8. doi: 10.1177/1479164111403334. PMID 21562061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment 2/05-10/06
Groups:
- Rosiglitazone: 4mg oral tablet once daily titrated to 8mg oral tablet once daily
- Placebo: blinded placebo treatment matching 4mg placebo tablet oral once daily titrated to 8mg matching placebo tablet oral once daily
Period: Overall Study
Arm/Group | Rosiglitazone | Placebo
Started | 74 | 76
Completed | 54 | 54
Not Completed | 20 | 22
Not completed — Withdrawal by Subject | 18 | 19
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone | Placebo | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 76 | 150
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 57.0 (8.7) | 55.7 (8.3) | 56.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 62
  Male | 42 | 46 | 88
Region of Enrollment [Number; unit: participants]
  United States | 74 | 76 | 150

OUTCOME MEASURES:

1. Secondary Outcome: Intra-myocardial Triglyceride Content Using in Vivo Magnetic Resonance Spectroscopy at 6 Months
Description: proton magnetic resonance spectroscopy determination of intra-myocardial triglyceride content at baseline and after 6 months, with triglyceride quantified analyzing fat and water signals assuming monoexponential signal decay and expressed as a percentage of fat-to-water (%)
Time Frame: 6 months
Population: analysis limited to those with interpretable imaging data at baseline and end of study
Measure: Mean (Standard Deviation); unit: percentage of fat-to-water; %
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 26 | 23
percentage of fat-to-water; % | 0.9 (0.49) | 0.85 (0.5)
Statistical Analysis 1: Comparison: Rosiglitazone vs Placebo; powered to detect at least 33% difference between groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

2. Primary Outcome: Peak Oxygen Uptake (VO2)
Description: measurement of peak oxygen uptake (VO2peak) during treadmill exercise, in units of milliliters of oxygen per kilogram of fat-free mass per minute
Time Frame: 6 months
Population: completed baseline and end-of-study cardiopulmonary exercise test
Measure: Mean (Standard Deviation); unit: ml O2 uptake/kg fat-free mass/minute
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 54 | 54
ml O2 uptake/kg fat-free mass/minute | 26.1 (7) | 27.6 (6.6)
Statistical Analysis 1: Comparison: Rosiglitazone vs Placebo; powered to detect difference of at least 10% between groups; Test type: Superiority or Other; p = 0.26, t-test, 2 sided

3. Secondary Outcome: Percentage of Patients Developing New or Worsening Peripheral Edema
Description: clinical evaluation of peripheral edema by physical exam at each study visit by a cardiologist using standard clinical severity scale 0-4, with new/worsening edema defined as any edema in patients with none at baseline, OR increase in severity by 2 or more points in patients with edema at baseline
Time Frame: 6 months
Measure: Number; unit: percentage of patients
Arm/Group | Rosiglitazone | Placebo
Number analyzed (Participants) | 74 | 76
percentage of patients | 54 | 33
Statistical Analysis 1: Comparison: Rosiglitazone vs Placebo; comparative incidence; Test type: Superiority or Other; p = 0.03, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Rosiglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 3/74 | 2/76
Other Adverse Events (participants affected / at risk) | 0/74 | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone (N=74) | Placebo (N=76)
heart failure (Cardiac disorders) | 3 (3) | 2 (2)
Heart failure (Cardiac disorders) | 3 (3) | 0 (0)
acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Larger than anticipated study discontinuation-72% with complete primary data analysis with lower numbers analyzed for imaging endpoints

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No